CLINICAL TRIAL: NCT01682486
Title: Evaluation of Tolerability, Safety and Performance of BIP Endotracheal Tubes With Bactiguard Coating
Brief Title: BIP ETT Clinical Tolerability, Safety and Performance Study
Acronym: BIPETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bactiguard AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1842-2026-CDOC
Record Dates: First submitted 2012-08-30; First posted 2012-09-11 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2014-07

CONDITIONS: Endotracheal Intubation During Surgery; Hospital Acquired Infections
Keywords: Medical device; Endotracheal Tube(s), ETT; Bactiguard Coated ETT; Tolerability; Safety; Performance; Bacterial colonization on ETT surface; Hospital Acquired Infections, HAI; Ventilator Associated Pneumonia, VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIP ETT, Bactigaurd coated endotracheal tube (Experimental)
  Interventions: Device: BIP ETT (Bactiguard)
- Standard ETT, un-coated endotracheal tube (Placebo Comparator)
  Interventions: Procedure: Standard ETT

INTERVENTIONS:
Device: BIP ETT (Bactiguard) — Ventilation of surgery patients during anesthesia using BIP ETT
  Other Names: BIP Endotracheal tube; Bactiguard coated ETT; Bactiguard coated Endotracheal tube
  Arms: BIP ETT, Bactigaurd coated endotracheal tube
Procedure: Standard ETT — Ventilation of surgery patients during anesthesia using standard ETT
  Other Names: ETT; Endotracheal tube; Standard Endotracheal tube; Uncoated ETT; Uncoated Endotracheal tube
  Arms: Standard ETT, un-coated endotracheal tube

SUMMARY:
The objective of the study is to determine Bactiguard coated BIP Endotracheal tube´s tolerability, safety and performance and compare it to a standard un-coated Endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* adult men and women >=18 years of age
* are, in opinion of the investigator able to communicate with and understand the trial personnel and comply with the requirements of the trial (e.g. fill in questionnaire)
* requiring endotracheal intubation >=3 h for elective surgery of upper gastrointestinal tract with a tube size of 7 or 8
* has signed informed consent

Exclusion Criteria:

* known transmissive blood disease
* known multiresistant bacterial colonization
* current and continuous treatment by immunomodulating therapies - e.g. systemic (or inhalation) use of cortisone or NSAIDS
* ongoing respiratory infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Tolerability assessment by using a symptom questionnaire (QLQ-H&N35) before and after surgery. Evaluation of tracheal mucosa directly during surgery and after the end of study by using photos. | Change from Baseline in symptoms and tracheal mucosa after surgery of expected average length of 5 hours

SECONDARY OUTCOMES:
Overall assessment of safety (device related adverse events and any problems in post postoperative course) | Participants will be followed on the surgery day and the day after surgery
Overall assessment of device performance | The performance will be followed during surgery of an expected average duration of 5 hours
  Recording of any device related problems experienced by the physician/health care personnel

OTHER OUTCOMES:
Develop a method for surrogate performance evaluation by microbial colonization testing of bacteria from the ETT surface | Microbial testing up to 1 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sigridur Kalman, MD PhD Prof, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bjorling G, Johansson D, Bergstrom L, Jalal S, Kohn I, Frostell C, Kalman S. Tolerability and performance of BIP endotracheal tubes with noble metal alloy coating--a randomized clinical evaluation study. BMC Anesthesiol. 2015 Dec 1;15:174. doi: 10.1186/s12871-015-0156-z. PMID 26625869